CLINICAL TRIAL: NCT00894179
Title: Feasibility, Safety and Accuracy of Regadenoson-Atropine ( REGAT) Stress Echocardiography for the Diagnosis of Coronary Artery Disease: An Angiographic Correlative Study
Brief Title: Safety and Accuracy Study of Regadenoson Atropine Combination for Stress Echocardiography in Identification of Coronary Artery Disease
Acronym: REGAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henry Ford Health System (Other)
Responsible Party: Karthikeyan Ananthasubramaniam, Henry Ford Hospital
Other Study IDs: REGA-9B04
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2010-05

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; stress echocardiography; regadenoson; atropine; coronary angiogram
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Purpose: The investigators plan to test a newly FDA approved pharmacologic stress agent, Regadenoson, in conjunction with atropine in the use of stress echocardiography for the diagnosis of coronary artery disease. The selective nature of Regadenoson allows for its use in patients with contraindications to the currently used drug, Adenosine, which is non-selective. Furthermore, the proposed protocol can be completed faster and without radiation exposure than the current protocol with adenosine.

Design: This is a prospective study evaluating people with no prior diagnosis of coronary disease with a prior stress test and are scheduled for cardiac catheterization. Patients who meet inclusion criteria will undergo regadenoson-atropine echocardiography protocol prior to their catheterization. The study will be interpreted by two independent readers blinded to the catheterization results. The sensitivity, specificity, positive and negative predictive values of the regadenoson-atropine study will be then be calculated using the coronary angiogram as a gold standard.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Able to provide consent
3. Scheduled for cardiac catheterization either with or without a prior functional stress imaging study

Exclusion Criteria:

1. Any history of acute myocardial infarction, prior PCI in last 3 months, bypass surgery,
2. History of greater than first degree AV block, sick sinus syndrome in patients
3. Patients with a pacemaker/LBBB
4. History on uncontrolled arrhythmias
5. Patients with significant pulmonary disease, known or suspected bronchoconstrictive or bronchospastic lung disease or other hypersensitivity to adenosine
6. History of cardiac transplantation, hypertrophic cardiomyopathy, acute myocarditis or pericarditis, severe valvular heart disease
7. Hemodynamically unstable patients
8. Dipyridamole use within 30 hours, consumption of methylxanthines (e.g., tea, coffee, caffeinated soft drinks, chocolate, or cocoa) within 12 hours, or use of sublingual nitroglycerin within 2 hours
9. History of glaucoma or obstructive uropathy
10. Allergy or hypersensitivity to atropine
11. Participation in another investigational drug study within 1 month or participation in any previous regadenoson trial
12. Pregnancy, breast feeding, or not using an acceptable method of birth control (if premenopausal)
13. . History of end-stage renal disease on hemodialysis or peritoneal dialysis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a prospective study evaluating stable outpatients with no prior diagnosis of coronary disease who may or may not have had a prior functional stress imaging test and are going for a clinically indicated cardiac catheterization as deemed by their physician due to suspected coronary artery disease either based on symptoms or based on results for prior functional testing
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2009-05; Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the sensitivity, specificity, positive and negative predictive value and accuracy of REGAT stress echocardiography protocol in the detection of coronary artery disease, using > 70% luminal stenosis on coronary angiogram as gold standard.

SECONDARY OUTCOMES:
Evaluate the safety and tolerability (using patient questionnaire) of REGAT stress echocardiography | 1-7 days after stress test
Compare sensitivity, specificity, positive and negative predicative value and accuracy of a REGAT stress echocardiography protocol to other stress imaging modalities used in the patient cohort as per design of study

CONTACTS AND LOCATIONS:
Overall Officials: Karthikeyan Ananthasubramaniam, MD FACC, Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States